CLINICAL TRIAL: NCT06299787
Title: Assessing the Role of Repetitive Transcranial Magnetic Stimulation on Aberrant Executive Function in the Context of Major Depressive Disorder in Adult Outpatients Seeking Treatment for Alcohol Use Disorder
Brief Title: Cognitive Dysfunction in the Addictions Study - Project 4 (P4)
Acronym: CDiA-P4
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 058-2021
Record Dates: First submitted 2022-10-13; First posted 2024-03-08 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Major Depressive Disorder; Alcohol Use Disorder
MeSH Terms: conditions — Depressive Disorder, Major; Alcoholism

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active Bilateral (Active Comparator): Bilteral TBS, applied as cTBS over the right DLPFC followed by iTBS over the left DLPFC
  Interventions: Device: intermittent theta burst stimulation
- Sham (Sham Comparator): Sham TBS
  Interventions: Device: Sham stimulation

INTERVENTIONS:
Device: intermittent theta burst stimulation — Theta-burst stimulation
  Arms: Active Bilateral
Device: Sham stimulation — Stimulation with double-sided B70-type coil
  Arms: Sham

SUMMARY:
The prefrontal cortex, although well established as an efficacious target for the treatment of major depressive disorder (MDD), has recently come into favour as a therapeutic target for alcohol use disorders (AUD). Depressive symptoms are also highly prevalent in individuals with AUD. A number of cognitive and psychological processes stemming from the prefrontal cortex, a common treatment target for repetitive transcranial magnetic stimulation (rTMS), are disrupted in both MDD and AUD. The proposed study will enhance the development of theta burst stimulation (TBS) as a new intervention for AUD in the context of depressive symptoms and uses integrated TMS-EEG to identify neurophysiological targets of executive dysfunction in this disorder.

DETAILED DESCRIPTION:
The prefrontal cortex, although well established as an efficacious target for the treatment of major depressive disorder (MDD), has recently come into favour as a therapeutic target for alcohol use disorders (AUD). Depressive symptoms are also highly prevalent in individuals with AUD. A number of cognitive and psychological processes stemming from the prefrontal cortex, a common treatment target for repetitive transcranial magnetic stimulation (rTMS), are disrupted in both MDD and AUD. The proposed study will enhance the development of theta burst stimulation (TBS) as a new intervention for AUD in the context of depressive symptoms and uses integrated TMS-EEG to identify neurophysiological targets of executive dysfunction in this disorder.

ELIGIBILITY:
Inclusion Criteria:

1. are outpatients;
2. are voluntary and competent to consent to treatment;
3. have a Diagnostic and Statistical Manual for Mental Disorders, 5th edition (DSM-5) diagnosis of AUD based on the MINI;
4. do not exhibit problematic use of any substances (excluding nicotine and caffeine), including alcohol, for >1 month;
5. are male or female between the ages of 18 - 59;
6. screened positive for an MDE based on the MINI without psychotic symptoms
7. are agreeable to keeping their current antidepressant medications and medications for alcohol use disorder constant during the study;
8. are reliably taking SUD agonist therapies if appropriate and managed by their clinical team;
9. are able to adhere to the study schedule;
10. meet the TMS safety criteria.

Exclusion Criteria:

1. have a concomitant major unstable medical illness;
2. are pregnant or intend to get pregnant during the study;
3. have possible or probable dementia (based on the Informant Questionnaire on Cognitive Decline in the Elderly that will be administered to any participant with a baseline total score of < 26 on the Montreal Cognitive Assessment (MoCA);
4. have failed a course of ECT, due to the lower likelihood of response to rTMS;
5. have any significant neurological disorder (e.g., a space occupying brain lesion, a history of stroke, a cerebral aneurysm, a seizure disorder, Parkinson's disease, Huntington's chorea, multiple sclerosis, significant history of head trauma with radiological evidence of intracranial trauma at the time of injury due to risk of possible seizure foci from prior intracranial lesions.
6. present with a medical condition, a medication, or a laboratory abnormality that could cause a major depressive episode or significant cognitive impairment in the opinion of the investigator (e.g., hypothyroidism with low TSH, Cushing's disease);
7. have an intracranial implant (e.g., aneurysm clips, shunts, cochlear implants) or any other metal object within or near the head, excluding the mouth, that cannot be safely removed;
8. require a benzodiazepine with a dose equivalent to lorazepam 2 mg/day or higher or any anticonvulsant due to the potential of these medications to limit the efficacy of rTMS [79];
9. have an inability to communicate in English fluently enough to complete the clinical assessments.
10. have a MINI diagnosis or active symptoms of Bipolar Disorder

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-02-07 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Executive Function Index - inhibition | baseline and 4 weeks after baseline (after 20 treatments of active/sham rTMS)
  Flanker task
Executive Function Index - working memory | baseline and 4 weeks after baseline (after 20 treatments of active/sham rTMS)
  N-back task
Executive Function Index - set shifting | baseline and 4 weeks after baseline (after 20 treatments of active/sham rTMS)
  switch task

SECONDARY OUTCOMES:
17-Item Hamilton Depression Rating Scale (HRSD-17) | baseline and 4 weeks after baseline (after 20 treatments of active/sham rTMS)
  Decrease in 17-Item Hamilton Depression Rating Scale score, 0 is lowest value, 52 is highest, higher value = more severe depression

OTHER OUTCOMES:
Columbia-Suicide Severity Rating Scale | baseline and 4 weeks after baseline (after 20 treatments of active/sham rTMS)
  Decrease in Columbia-Suicide Severity Rating Scale score, 0 is lowest score, 25 is highest, higher value = more suicidal ideation

CONTACTS AND LOCATIONS:
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada